CLINICAL TRIAL: NCT07326943
Title: Minimum Effective Dose of Ropivacaine 0.5% for Ultrasound-guided Interscalene Block Targeting the C7 Nerve Root in Hand and Forearm Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua Zheng, Head of the Anesthesiology Department, Huazhong University of Science and Technology
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: YXLL-2025-292
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Intermuscular Groove Brachial Plexus Block
Keywords: ultrasound-guided interscalene block; Minimum effective dose; C7 nerve root

STUDY DESIGN:
Intervention Model Description: This experiment enrolled participants using a biased coin up and down sequential method. The first subject was given 0.5% ropivacaine 12mL. The subsequent dose of ropivacaine for each subject depends on the anesthetic effect of the previous subject. If the effect of the previous subject is "failure" (negative reaction), the dose of ropivacaine will be increased by 1mL for the next subject. If the effect of the previous subject is "success" (positive reaction), the next subject will be randomized using the partial currency method. The patients will be randomly divided into two groups: one group will receive the same dose of ropivacaine as the previous subject (probability B=0.89) (same dose group); The dose of ropivacaine in another group decreased by 1mL (probability 1-B=0.11). The criterion for successful blockade is to simultaneously meet the following two criteria: (1) disappearance of sensory sensation in the muscle cutaneous nerve, medial forearm cutaneous nerve, median nerve, rad
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deceasing (Experimental): Brachial plexus block with decreasing dose. Real time ultrasound-guided intermuscular brachial plexus block anesthesia targeting the C7 nerve root.
  Interventions: Procedure: Ultrasound guided intermuscular groove block
- similar (Experimental): Brachial plexus block, with similar doses. Real time ultrasound-guided intermuscular brachial plexus block anesthesia for C7 nerve roots
  Interventions: Procedure: Ultrasound guided intermuscular groove block

INTERVENTIONS:
Procedure: Ultrasound guided intermuscular groove block — The patient will receive ultrasound-guided intermuscular groove brachial plexus block targeting the C7 nerve root, decreasing doses of ropivacaine 0.5% will be administered.
  Arms: Deceasing
Procedure: Ultrasound guided intermuscular groove block — The patient will receive ultrasound-guided intermuscular groove brachial plexus block targeting the C7 nerve root, similar doses of ropivacaine 0.5% will be administered.
  Arms: similar

SUMMARY:
Inter muscular groove brachial plexus block is a commonly used peripheral nerve block technique in clinical practice, commonly used for anesthesia and analgesia in clavicle, shoulder, and humeral surgeries. Intermuscular groove block is achieved by injecting local anesthetics between the anterior and middle scalene muscles in order to block the anterior branches of the cervical nerve that pass through this gap, including the anterior branches of the cervical 5 (C5), cervical 6 (C6), and cervical 7 (C7) spinal nerves. The classic technique of intermuscular groove block involves puncturing the thyroid cartilage horizontally into the intermuscular groove. This area is roughly equivalent to the level of the anterior branch of the C5/C6 nerve root. The classic ultrasound-guided intermuscular groove block also involves puncturing the needle to the level of the C5/C6 anterior branch for drug injection. After injection, local anesthetics mainly wrap around C5, C6, and some C7 nerve roots. According to the range of spinal nerve innervation, its blocking range is located in the shoulder, the anterior, posterior, and lateral sides of the upper arm, the anterior, posterior, and lateral sides of the forearm, and the two and a half fingers on the radial side. Therefore, intermuscular groove block is mainly used for shoulder, humerus, and clavicle surgery. Due to incomplete ulnar block, it is not recommended for surgery on the elbow joint and its distal end.

Scholars have found that using C5 as the puncture target to implement intermuscular groove block and administering 10ml of 0.75% ropivacaine, the success rate of ulnar nerve block is 19%. The success rate of ulnar nerve block with C6 as the puncture target was 93% when 10ml of 0.75% ropivacaine was administered. This suggests that blockade methods closer to the tail muscle groove on the tail side have a higher success rate for blocking the C7, C8, and T1 nerve roots. In our clinical work, we found that when performing intermuscular groove block with C7 nerve root as the puncture target, local anesthetics not only stably wrap around C7 nerve root, but also spread to wrap around C5 and C6 nerve roots on the head side, and spread to the deep surface of the brachial plexus trunk on the tail side. Local anesthetic diffusion can also be seen in some patients at the brachial plexus bundle in the intercostal space. From the perspective of local anesthetic diffusion patterns, intermuscular groove block targeting the C7 nerve root may cover the anterior branches of C5, C6, C7, C8, and T1 nerve roots, achieving complete brachial plexus block. In the preliminary exploratory clinical work, the patient underwent C7 nerve root intermuscular groove brachial plexus block. Through sensory testing, it was found that the musculocutaneous nerve, medial forearm nerve, radial nerve, median nerve, and ulnar nerve could all be stably blocked, and the forearm and hand surgeries were successfully completed under nerve block. Preliminary clinical practice suggests that C7 intermuscular groove block can be used for forearm and hand surgery. Successful C7 intermuscular groove block relies on the diffusion and wrapping of local anesthetics around the anterior branches of C5, C6, and C7 nerve roots, as well as the inferior trunk of the brachial plexus (or the anterior branches of C8 and T1 nerve roots).

Therefore, we designed this study to determine the amount of local anesthetic required to achieve stable forearm and hand block during C7 intermuscular groove block.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age range: 18-60 years old (2) ASAⅠ~II (3) BMI between 18 and 30kg/m2 (4) Patients undergoing hand or forearm surgery (5) Sign informed consent form

Exclusion Criteria:

* (1) Refusal to participate in the experiment (2) Merge peripheral nerve diseases (3) Lidocaine and ropivacaine allergy (4) Pregnant women (5) Obstructive or restrictive lung disease (6) Coagulation dysfunction (7) Long term use of opioid drugs (8) Infection, tumor or surgical history at the puncture site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of blocking effect | From the completion of nerve block to the 30th minute after block
  Starting from the completion of the nerve block, an independent evaluator (unaware of the dosage used) will test and record the block effect at 10, 20, and 30 minutes after the block. The block effect will be judged based on the effect at 30 minutes. Conduct sensory tests on the skin innervated by various nerves using ice cubes. Use a 3-point numerical scale (0=normal cold sensation, no obstruction; 1=partial cold sensation, partial obstruction; 2=no cold sensation, complete obstruction). Radial nerve, median nerve, ulnar nerve, musculocutaneous nerve, and medial forearm cutaneous nerve. Evaluate the degree of motor block through specific exercise activities (0=normal activity, 1=partial block, 2=complete block). Patients who are fully awake or have been administered an appropriate amount of sedatives, maintain spontaneous breathing, and successfully complete the surgery are considered to have successful blockade (i.e. positive reaction).

SECONDARY OUTCOMES:
Diaphragmatic muscle movement status | From the completion of nerve block to the 30th minute after block
  Ultrasound measurement of basal range of motion of the blocked ipsilateral diaphragm: The patient is seated in a semi seated position, with a low-frequency convex array probe placed between the anterior axillary line and the midline of the axilla. Real time M-mode ultrasound is used to evaluate the motion of the ipsilateral diaphragm. Use a low intercostal or subcostal approach, with the liver or spleen as the sound window for scanning. Record the diaphragm movement amplitude during rapid nasal inhalation from the resting exhalation position. Measure three times and take the average. And retain the measured images.
  30 minutes after the completion of nerve block, evaluate the patient's diaphragm movement using the same method as before. The degree of diaphragmatic block is defined as a decrease in movement amplitude of>75% (complete diaphragmatic block), a decrease in movement amplitude of 25-75% (partial block), and a decrease of<25% (no block) compared to before the block was impleme

OTHER OUTCOMES:
Complications of nerve block | From the completion of nerve block to the 30th minute after block
  The evaluator also records the occurrence of complications such as hypersensitivity, vascular injury, recurrent laryngeal nerve block, Horner's syndrome, and local anesthetic poisoning during the blocking process.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
Paper case report forms were written by hand